CLINICAL TRIAL: NCT00001659
Title: Conjugal Bereavement in Older Adults: Biological, Functional, and Psychological Consequences
Brief Title: Consequences of Conjugal Bereavement in Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970157; 97-M-0157
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-05

CONDITIONS: Bereavement; Depressive Disorder; Immunologic Disease; Mental Disorder; Sleep Disorder
Keywords: Bereavement; Depression; Suicide; Activity of Daily Living; Immune Function; Occupational Performance; Sleep Disorders; Mood Changes
MeSH Terms: conditions — Depressive Disorder; Immune System Diseases; Mental Disorders; Sleep Wake Disorders; Depression; Suicide

SUMMARY:
Bereavement refers to the expected reactions and sadness associated with the loss of a loved one. It has been reported that the loss of a spouse is rated as the major life stressor among survivors of varying ages and diverse cultural backgrounds. Statistics have shown that in the United States over 800,000 men and women lose a spouse each year.

A wide range of symptoms has been associated with bereavement including; depressed mood, tearfulness, sleep disturbances, and irrational behavior. Previous studies have shown that up to 50% of bereaved individuals can develop major depression. Bereavement has also been associated with dysfunction of the immune system. As a result, bereaved adults are more vulnerable to infection. However, the exact relationship between bereavement and immunity is uncertain.

Researchers firmly believe that a relationship does exist between stress, more specifically bereavement, immunity, and the increased chance of dying following the loss of a long-term spouse.

The objective of this study is to find possible links between bereavement, depression, and the immune system. This study will follow a group of elderly bereaved spouses and a group of elderly people who have not lost a long-term spouse. The group of bereaved individuals will be followed for approximately 13 months after the loss of their spouse and the group of controls will be followed for 13 months after entering the study. Researchers will make note of any clinical, biological, and immunological changes in any participants of the study.

DETAILED DESCRIPTION:
It is estimated that over 800,000 men and women become bereaved each year in the United States (LaRue et al, 1985). While the near certainty of such bereavement is predictable in one spouse or the other, the exact impact and duration of bereavement is much less predictable (Stroebe et al, 1995). It has been reported that the loss of a spouse is rated as the major life stressor among survivors of varying ages and diverse cultural backgrounds (Holmes and Rahe, 1967). As one copes with the loss of a loved one, expected reactions include sadness, tearfulness, and even depression (DeLeon, 1994; Pasternak, 1996). Other complications can include work-related difficulties, sleep disturbances, irrational behaviors, and immunologic dysfunction (Zisook, 1994; Prigerson, et al, 1995). All of these symptoms are common; yet, the underlying biology and relationship with the time course of bereavement are still poorly understood. The purpose of this study will be to prospectively follow a cohort of elderly bereaved spouses and controls from multiple clinical and biological perspectives over thirteen months after the loss of a spouse.

ELIGIBILITY:
People over the age of 50 who have lost their spouse within the last three months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Start 1997-07; Study Completion 2002-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kiecolt-Glaser JK, Glaser R, Gravenstein S, Malarkey WB, Sheridan J. Chronic stress alters the immune response to influenza virus vaccine in older adults. Proc Natl Acad Sci U S A. 1996 Apr 2;93(7):3043-7. doi: 10.1073/pnas.93.7.3043. PMID 8610165
- [Background] Reynolds CF 3rd, Frank E, Perel JM, Mazumdar S, Kupfer DJ. Maintenance therapies for late-life recurrent major depression: research and review circa 1995. Int Psychogeriatr. 1995;7 Suppl:27-39. doi: 10.1017/s104161029500233x. PMID 8580390
- [Background] Steffens DC, Plassman BL, Helms MJ, Welsh-Bohmer KA, Saunders AM, Breitner JC. A twin study of late-onset depression and apolipoprotein E epsilon 4 as risk factors for Alzheimer's disease. Biol Psychiatry. 1997 Apr 15;41(8):851-6. doi: 10.1016/S0006-3223(96)00247-8. PMID 9099411